CLINICAL TRIAL: NCT02517541
Title: A Clinical Investigation Evaluating and Understanding Parameters Affecting the Performance of Ostomy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP259
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Ileostomy - Stoma; Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test period (Experimental): The arm consists of a two-week baseline period where subjects apply their own product and a 12 weeks test period where the subjects apply the intervention (SenSura Mio Convex Soft)
  Interventions: Device: SenSura Mio Convex Soft

INTERVENTIONS:
Device: SenSura Mio Convex Soft — SenSura Mio Convex Soft is a CE marked ostomy product manufactured by Coloplast

SUMMARY:
The aim of the study is to obtain an understanding of relevant parameters affecting the performance of ostomy products.

DETAILED DESCRIPTION:
72 subjects will be included. Each subject will attend 3 visits at the clinic/hospital or at the subjects home depending on the final site set-up. Each subject will be enrolled for 14 weeks in total for the entire investigation.

Coloplast will provide SenSura Mio Convex Soft for all subjects via the investigator. Based on the subjects' usual changing pattern, the investigator will provide the subjects with enough products for the whole test period.

The subject will answer questions regarding the tested products by filling out the subject part in the eCRF daily. The subject will answer questions using an electronic device and use the device to take pictures of the peristomal skin and used products at each product change. The Investigator fills out the investigator part of the eCRF at each visit. The subjects must complete the general questions at the end of each test period before their second and third visit at the Clinic/hospital or at home to avoid influence by the investigator.

The use of accessories will be noted in the eCRF. Samples of biological material will not be taken or used in this investigation. Patient files from own physician will not be used for subjects recruited via a Coloplast's database. The investigators may use patient files for subjects recruited via hospital sites/ostomy clinics to identifying relevant subjects and/or to verify baseline information, concomitant medication or adverse events. To be able to fulfil the objectives, the investigation must include both ileostomists and colostomists.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have an ileostomy or colostomy
* Have had their ostomy for at least 3 months
* Must use 1 piece open or closed ostomy products during the test period
* Currently using a 1 piece. flat product
* Must be able to use custom cut product
* Have intact peristomal skin
* Has experienced leakage (seeping) under the baseplate at least three times during the last two weeks
* Are evaluated to be suitable for a soft convex product

Exclusion Criteria:

* Currently receiving or have within the past 2 month received radio- and/or chemotherapy
* Currently or having within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
* Are pregnant or breastfeeding
* Participating in other interventional clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla F Vibjerg, M.Sc.pharm, Study Chair — Head of Clinical Operations
Locations (9):
- United States (2):
  - University of Chicago Medicine, Chicago, Illinois
  - Prism research center, Saint Paul, Minnesota
- QPS Netherlands, Groningen, Netherlands
- Helse Nordbyen, Larvik, Norway
- United Kingdom (5):
  - Synexus Midlands, Birmingham
  - Pilgrim Hospital, Boston
  - Cheltenham General Hospital, Cheltenham
  - Kettering General hospital, Kettering
  - Lincon Country hospital, Lincoln

RESULTS

PARTICIPANT FLOW:
Period: Baseline Period (Own Product)
Arm/Group | Test Period
Started | 74
Completed | 73
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Test Period (SenSura Mio Convex Soft)
Arm/Group | Test Period
Started | 73
Completed | 61
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — One subjects was not suited for the tes | 2

BASELINE CHARACTERISTICS:
Population: All subjects who were included in the safety population of the investigation. One subject did not provide baseline data as the subject violated the protocol and terminated the study. Therefore, no baseline data was recorded.
Arm/Group | Test Period
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Leakage Under the Baseplate (cm^2)
Description: The leakage area was measured using photos of used baseplates. A computer program was used to measure the leakage area.
Time Frame: 14 weeks (2 weeks baseline + 12 weeks intervention)
Measure: Mean (Standard Deviation); unit: cm2
Units Other Than Participants: baseplates
Groups:
- Own Product: The mean leakage area measured on the subjects own baseplate
- SenSura Mio Convex Soft: The mean leakage area measured on SenSura Mio Convex Soft baseplates
Arm/Group | Own Product | SenSura Mio Convex Soft
Number analyzed (Participants) | 73 | 73
Number analyzed (baseplates) | 925 | 796
cm2 | 9.2 (9.8) | 6.6 (8.2)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in the study period (14 weeks)
Arm/Group | Own Product | SenSura Mio Convex Soft
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/71
Other Adverse Events (participants affected / at risk) | 17/74 | 25/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Own Product (N=74) | SenSura Mio Convex Soft (N=71)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — During a routine visit at the hospital her potassium values were too low so the medical staff decided to keep her overnight and administer potassium by means of an IV drip
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Own Product (N=74) | SenSura Mio Convex Soft (N=71)
Peristomal skin dermatitis (Skin and subcutaneous tissue disorders) | 17 (20) | 25 (59) — Red, eroded peristomal skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less